CLINICAL TRIAL: NCT05603650
Title: Effects of Mouthrinses on the Microbiome of the Oral Cavity and GI Tract
Brief Title: Effects of Mouthrinse on the Microbiome of the Oral Cavity and GI Tract
Acronym: Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Petra E. Wilder-Smith, Professor of Surgery and Director of Dentistry, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20205719
Record Dates: First submitted 2022-09-12; First posted 2022-11-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Oral Bacterial Infection; Oral Infection; Microbial Colonization; Viral Infection
Keywords: Oral Microbiome; Fecal Microbiome
MeSH Terms: conditions — Communicable Diseases; Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: White tape over receptacle
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water rinse (Placebo Comparator): rinse twice daily for 1 min with water
  Interventions: Other: Lumineux Oral Essentials rinse; Other: Listerine rinse
- Lumineux Oral Essentials rinse (Experimental): rinse twice daily for 1 min with Lumineux Oral Essentials rinse
  Interventions: Other: Listerine rinse
- Listerine rinse (Experimental): rinse twice daily for 1 min with Listerine rinse
  Interventions: Other: Lumineux Oral Essentials rinse

INTERVENTIONS:
Other: Lumineux Oral Essentials rinse — mouthrinse
  Arms: Listerine rinse; Water rinse
Other: Listerine rinse — mouthrinse
  Arms: Lumineux Oral Essentials rinse; Water rinse

SUMMARY:
The purpose of this research study is to identify the effects of 2 over-the-counter mouthwashes on bacteria and 3 viruses in the participant's mouth and gut. The participant will be randomly allocated to rinse their mouth twice daily either with Listerine mouthwash, Lumineux Oral Essentials mouthwash, or water. The overall duration of the study will be approximately 180 days and will include approximately 5 visits and 15-30 minutes for each visit with a total of approximately 2.5 hours of your time. Additionally, fecal matter will also be collected in some subjects using a commercial collection kit.

DETAILED DESCRIPTION:
Goal of this pilot study is to identify the effects of 2 over-the-counter mouthrinses on the microbiome of the oral cavity and the GI tract. We will investigate 2 mouthwashes, plus an additional non-treatment group (water rinse only). One mouthwash has antimicrobial activity (ListerineR, Johnson & Johnson Consumer Healthcare Products, Skillman, New Jersey); the other targets microbial products only (Lumineux Oral Essentials Clean and Fresh MouthwashR, Los Angeles, CA). Oral plaque will be collected with a sterile swab using a commercial collection kit on Day 0, Day 30, Day 60, Day 90, and Day 180 of the study. Additionally, fecal matter will also be collected in some subjects using a commercial collection kit. Subjects will rinse 2x daily for approximately 180 days using either mouthwash or water.

ELIGIBILITY:
Inclusion Criteria:

* Eligible men and non-pregnant and non-lactating women of all races age 18-25.
* Volunteers must consent to participate in all scheduled exam visits and procedures.
* Volunteers must be available for follow up on the telephone.
* Healthy gums or gums that bleed when you brush them.

Exclusion Criteria:

* Volunteers unable or unwilling to sign the informed consent form.
* Less than 20 teeth (excluding third molars).
* Individuals who have taken antibiotics in the previous 3 months.
* Presence of any condition, abnormality, or situation at Baseline that in the opinion of the Principal Investigator may preclude the volunteer's ability to comply with study requirements, including completion of the study or the quality of the data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
total bacterial load and mRNA analysis | Day 0
  total bacterial load as determined from oral swabs and collected fecal samples, followed by subsequent standard mRNA analysis using RT-PCR
total bacterial load and mRNA analysis | Day 30
  total bacterial load as determined from oral swabs and collected fecal samples, followed by subsequent standard mRNA analysis using RT-PCR
total bacterial load and mRNA analysis | Day 60
  total bacterial load as determined from oral swabs and collected fecal samples, followed by subsequent standard mRNA analysis using RT-PCR
total bacterial load and mRNA analysis | Day 90
  total bacterial load as determined from oral swabs and collected fecal samples, followed by subsequent standard mRNA analysis using RT-PCR
total bacterial load and mRNA analysis | Day 180
  total bacterial load as determined from oral swabs and collected fecal samples, followed by subsequent standard mRNA analysis using RT-PCR
viral load and mRNA analysis using RT-PCR | Day 0
  viral load: HSV1, CMV, EBV
viral load and mRNA analysis using RT-PCR | Day 30
  viral load: HSV1, CMV, EBV
viral load and mRNA analysis using RT-PCR | Day 60
  viral load: HSV1, CMV, EBV
viral load and mRNA analysis using RT-PCR | Day 90
  viral load: HSV1, CMV, EBV
viral load and mRNA analysis using RT-PCR | Day 180
  viral load: HSV1, CMV, EBV

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wilder-Smith, DDS, PhD, Principal Investigator — University of Calfornia Irvine
Locations (1):
- Beckman Laser Institute and Medical Clinic, Irvine, California, United States